CLINICAL TRIAL: NCT02009813
Title: Hyperbaric Oxygen Therapy and Insulin Resistance (HOTAIR2) - Effect of One HBO Session.
Acronym: HOTAIR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, A/Prof, University of Adelaide
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RAH121212a
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Insulin resistance; Inflammation; Hypoxia
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation; Hypoxia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — Participants will undergo 2 treatments of hyperbaric oxygen. Each treatment consists of 90 minutes compression at 2 atmospheres of pressure, with 30 minutes decompression back to 1 atmosphere. During this time, patients will be treated with 100% oxygen delivered via a hood system.

SUMMARY:
Obesity is an epidemic in Western society and is the biggest risk factor for insulin resistance and type 2 diabetes. The investigators have recently shown that exposure to hyperbaric oxygen (HBO) leads to an increase insulin sensitivity in males ubjects and that this improvement can be measured in all men, not just those with diabetes. The aim of this study is to investigate the time course of this effect and explore the mechanisms involved. The investigators suspect that insulin sensitivity as measured by hyperinsulinaemic-euglycaemic clamp will be increased within the time-frame of one 2-hour hyperbaric oxygen exposure, and that the improvement will be measurable in females as well as males.

ELIGIBILITY:
Inclusion Criteria:

* Overweight to obese (BMI 25-35 kg/m2)
* Age >18 years (no specific upper age limit)
* Fit to enter hyperbaric chamber as assessed by hyperbaric physician.

Exclusion Criteria:

* Personal history of Diabetes
* Personal history of major psychiatric disorders
* UIse of prescribed or non-prescribed medications which may affect glucose homeostasis (e.g. steroids),
* Uncontrolled asthma,
* Current fever or upper respiratory infections
* Individuals who regularly perform high intensity exercise (>2 week),
* Pregnancy, lactation and women who are planning to become pregnant
* Current intake of >140g alcohol/week,
* Current smokers of cigarettes/cigars/marijuana,
* Current inatke of any illicit substance,
* Claustrophobia
* has donated blood within past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 hours

SECONDARY OUTCOMES:
Hypoxia and inflammatory markers | 2 hours
  Using immuno-histo chemistry (IHC), quantitative plymerase chain reaction (qPCR), Western blot

CONTACTS AND LOCATIONS:
Overall Officials: Leonie K Heilbronn, PhD, Principal Investigator — University of Adelaide; David Wilkinson, BMBS, Principal Investigator — University of Adelaide
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Chen M, Liu B, Wilkinson D, Hutchison AT, Thompson CH, Wittert GA, Heilbronn LK. Selenoprotein P is elevated in individuals with obesity, but is not independently associated with insulin resistance. Obes Res Clin Pract. 2017 Mar-Apr;11(2):227-232. doi: 10.1016/j.orcp.2016.07.004. Epub 2016 Aug 11. PMID 27524654